CLINICAL TRIAL: NCT00593749
Title: Healthy Corner Store Initiative
Acronym: HCSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NEP - 10520; 10520
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2008-01

CONDITIONS: Obesity Prevention
Keywords: obesity prevention; corner stores; schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCS (Active Comparator): Intervention group
  Interventions: Behavioral: Healthy Corner Store Initiative
- Control (Placebo Comparator): Control
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Healthy Corner Store Initiative — modification of snacks and beverages offered in corner store surrounding 10 schools
  Other Names: HCSI
  Arms: HCS
Behavioral: Control — control group in study
  Arms: Control

SUMMARY:
The proposed research will evaluate the efficacy of an intervention in urban corner stores. Community-based, environmental manipulation of corner stores is an understudied area and represents the next step in understanding and improving the nutritional intake of school students to prevent obesity.

DETAILED DESCRIPTION:
The HCSI is a community-based, multi-faceted, and broad-based intervention administered by The Food Trust. The HCSI is designed to permeate multiple aspects (i.e., social, educational, food availability) of the corner store environment. Moreover, it takes into account the unique aspects of each corner store.

Theoretical Framework. The HCSI is grounded in social cognitive theory (SCT). By incorporating the environment, personal factors (including cognitions) and behavior, SCT provides a framework for designing, implementing, and evaluating behavioral change. It supports traditional behavioral methods (positive reinforcement, specific behavioral outcomes). Moreover, it underscores the critical role of the social environment (modeling, social reinforcement, social norms - as well as reducing the antecedents for purchasing unhealthy foods) in affecting change. Our initial work has assessed the feasibility of implementing the HCSI and collecting data (see preliminary studies). We are poised to test the efficacy of the HCSI in the proposed study.

Behavioral Goals. The HCSI intervention seeks to: 1) decrease the purchase of high calorie snacks and beverages and to 2) increase the percentage of healthy snacks and beverages at the store level. Decreasing the purchase of high-calorie foods in the corner stores and/or decreasing sugar-sweetened soft drinks (assuming no change in physical activity) will shift energy balance to favor the prevention of overweight and obesity. These dietary goals are also consistent with the Institute of Medicine report on childhood obesity (Preventing Childhood Obesity: Health in the Balance, 2004). While we will measure BMI in the proposed study, our primary outcome of this initial randomized trial of efficacy is energy intake assessed at the time of purchase.

Although the implementation of the intervention will vary depending on the characteristics of the corner store, the major components of the program are summarized below:

Key informant interviews with corner store owners and teachers at local schools and after-school programs to determine how best to work with these key groups Social marketing campaign to reinforce messages about healthy snacking, Grouping healthy snacks and/or displaying signage for easy identification of healthier items, Integrating healthy snacking information into school and after-school programs to teach youngsters what comprises a healthy snack Involving family members and the community in promoting healthy snacking Working with snack and beverage manufacturers and distributors to increase the number of healthy snacks available in corner stores.

ELIGIBILITY:
Inclusion Criteria:

* 4th, 5th and 6th grade students
* Schools who meet eligibility for 50% of students eligible to receive free or reduced lunches at their school
* Corner stores surrounding these schools within a 4 block radius in either direction

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To compare the intervention and control on changes, over a 2 year period, in the energy content of snacks purchased before and after school at corner stores. | post

SECONDARY OUTCOMES:
To compare the intervention and control groups on the percentage of available healthy snacks, the percentage of dedicated space for shelving healthy snacks, and the allocation of dedicated space where healthy items will be grouped for display. | post
To understand the correlates and determinants of corner store shopping behavior. | post

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — Temple University- Center for Obesity Research and Education
Locations (1):
- Temple University - Center for Obesity Research and Education, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Borradaile KE, Sherman S, Vander Veur SS, McCoy T, Sandoval B, Nachmani J, Karpyn A, Foster GD. Snacking in children: the role of urban corner stores. Pediatrics. 2009 Nov;124(5):1293-8. doi: 10.1542/peds.2009-0964. Epub 2009 Oct 12. PMID 19822591